CLINICAL TRIAL: NCT03596892
Title: Decitabine+Busulfan+Cyclophosphamide vs Busulfan+Cyclophosphamide Conditioning Regimen for Mixed-lineage-leukemia (MLL)-Rearranged Acute Leukemia Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Decitabine+BUCY vs BUCY Conditioning Regimen for MLL+ Acute Leukemia Undergoing Allo-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Peking University People's Hospital (Other); Zhujiang Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dec+BUCYvsBUCY-MLL+ AL-2018
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation; Conditions; Mixed-lineage-leukemia (MLL)-Rearranged Acute Leukemia
MeSH Terms: conditions — Disease | interventions — Decitabine; Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decitabine + BUCY (Experimental): For MLL+ acute leukemia undergoing allo-HSCT，Decitabine+BUCY conditioning regimen was Decitabine 20mg/m2/day on days -14 and -10； Busulfan (BU) 3.2 mg/kg/day on days -7 and -4；Cyclophosphamide (CY) 60 mg/kg/day on days -3 and -2.
  Interventions: Drug: Decitabine; Drug: Busulfan (BU); Drug: Cyclophosphamide (CY)
- BUCY (Active Comparator): For MLL+ acute leukemia undergoing allo-HSCT，BUCY conditioning regimen was Busulfan (BU) 3.2 mg/kg/day on days -7 and -4；Cyclophosphamide (CY) 60 mg/kg/day on days -3 and -2.
  Interventions: Drug: Busulfan (BU); Drug: Cyclophosphamide (CY)

INTERVENTIONS:
Drug: Decitabine — Decitabine was administered at 20mg/m2/day on days -14 and -10.
  Arms: Decitabine + BUCY
Drug: Busulfan (BU) — Busulfan was administered at 3.2 mg/kg/day on days -7 to -4.
Drug: Cyclophosphamide (CY) — Cyclophosphamide was administered at 60 mg/kg/day on days -3 to -2.

SUMMARY:
Recent studies demonstrated that allogeneic hematopoietic stem cell transplantation (allo-HSCT) could be a valuable treatment choice for mixed-lineage-leukemia (MLL)-rearranged acute leukemia. Unfortunately, some patients relapsed after allo-HSCT. In this prospective randomized controlled study, the safety and efficacy of Decitabine + BUCY and BUCY myeloablative conditioning regimens in MLL+ acute leukemia undergoing allo-HSCT are evaluated.

DETAILED DESCRIPTION:
Recent studies demonstrated that allogeneic hematopoietic stem cell transplantation (allo-HSCT) could be a valuable treatment choice for mixed-lineage-leukemia (MLL)-rearranged acute leukemia. BUCY conditioning regimen is the standard myeloablative regimen for MLL+ acute leukemia undergoing allo-HSCT. However, it appears to have higher relapse rate and lower survival. To reduce the relapse rate and improve the survival, decitabine is added in the conditioning regimen. In this prospective randomized controlled study, the safety and efficacy of Decitabine + BUCY and BUCY myeloablative conditioning regimens in MLL+ acute leukemia undergoing allo-HSCT are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* MLL+ acute leukemia undergoing allo-HSCT
* 14-65 years

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
relapse rate | 2 year

SECONDARY OUTCOMES:
overall survival (OS) | 2 year
disease-free survival (DFS) | 2 year
transplant-related mortality (TRM) | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China